CLINICAL TRIAL: NCT03414229
Title: Phase II Study of Epacadostat (INCB024360) in Combination With Pembrolizumab in Patients With Locally Advanced/Metastatic Sarcoma
Brief Title: A Study of Epacadostat, an IDO1 Inhibitor, in Combination With Pembrolizumab in Patients With Metastatic and/or Locally Advanced Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Incyte Corporation (Industry); Merck Sharp & Dohme LLC (Industry); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-508
Record Dates: First submitted 2018-01-23; First posted 2018-01-29 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Sarcoma
Keywords: Epacadostat; Pembrolizumab; 17-508
MeSH Terms: conditions — Sarcoma | interventions — epacadostat; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a single-center, phase II study to evaluate the efficacy of the IDO1 inhibitor, epacadostat, given in combination with the anti-PD1 monoclonal antibody, pembrolizumab, for patients with metastatic and/or locally advanced grade sarcomas.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- UPS, Liposarcoma or pleomorphic liposarcoma (Experimental): Undifferentiated Pleomorphic Sarcoma (UPS) or Liposarcoma (dedifferentiated or pleomorphic liposarcoma) Epacadostat 100mg Twice daily Continuously days 1-21 of each 3 week cycle Oral Pembrolizumab 200mg Every 3 weeks Day 1 of each 3 week cycle IV infusion
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab
- Leiomyosarcoma (Experimental): Epacadostat 100mg Twice daily Continuously days 1-21 of each 3 week cycle Oral Pembrolizumab 200mg Every 3 weeks Day 1 of each 3 week cycle IV infusion
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab
- Vascular Sarcoma Subtypes (Experimental): Including angiosarcoma and Epithelioid Hemangioendothelioma (EHE). Epacadostat 100mg Twice daily Continuously days 1-21 of each 3 week cycle Oral Pembrolizumab 200mg Every 3 weeks Day 1 of each 3 week cycle IV infusion
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab
- Other (Experimental): Epacadostat 100mg Twice daily Continuously days 1-21 of each 3 week cycle Oral Pembrolizumab 200mg Every 3 weeks Day 1 of each 3 week cycle IV infusion
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Epacadostat — 100mg bid days 1-21
Drug: Pembrolizumab — 200mg/dose Day 1, Q 3 weeks

SUMMARY:
The purpose of this study is to test any good and bad effects of the combination therapy of epacadostat and pembrolizumab and to determine how well the combination therapy works in the treatment of patients with sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years at the time of informed consent
* Be willing and able to provide written informed consent/assent for the trial
* Be willing to comply with treatment protocol
* Subjects must have a histologically confirmed metastatic and/or locally advanced sarcoma
* Adequate performance status: ECOG 0 or 1/KPS 100-70%
* Subjects must have at least one prior line of systemic therapy (e.g. chemotherapy, immunotherapy, targeted or biological therapy) for their sarcoma. An exception to this criterion will be made for patients with sarcoma histological subtypes for which there is no known standard systemic therapy (e.g., chondrosarcoma). Any patient that refuses standard chemotherapy for the treatment of their disease is also considered eligible. Prior adjuvant therapy will not count provided it was completed more than 6 months previously.
* Presence of measureable disease per RECIST v1.1.Target lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment.
* All subjects must agree to pre-treatment tumor biopsy. Subjects in whom biopsy is technically not feasible or in whom would result in unacceptable risk, in the opinion of the investigator, may be exempted from the biopsy requirement with discussion with the principal investigator.
* Adequate organ function determined within 21 days of treatment initiation
* Hematological

  * Absolute neutrophil count (ANC) ≥1,000 /mcL
  * Platelets ≥75,000 / mcL
  * Hemoglobin ≥8 g/dL or ≥5.0 mmol/L
* Renal

  °Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR

  ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN aCreatinine clearance should be calculated per institutional standard.
* Hepatic

  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin ≥ 2.5 mg/dL
* Coagulation

  * International Normalized Ratio 52 or Prothrombin Time ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Women of childbearing potential must have a negative serum pregnancy test at screening and ≤ 72 hours prior to day 1 of study treatment.
* Male and female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 11.7, for the course of the study through 120 days after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Uncontrolled intercurrent illness including current active infection requiring systemic therapy or symptomatic congestive heart failure within 6 months
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to enrollment. However, in the setting of non-immune mediated indications for steroid use, chronic/active low dose steroid use may be permitted at the discretion of the principal investigator. The dose of steroid allowed in this setting is also at the discretion of the principal investigator. (Use of inhaled or topical steroids is permitted.)
* History or evidence of symptomatic autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 years prior to enrollment. Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease.
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) disease
* Has known active Hepatitis B (e.g., Hepatitis B Virus PCR is detected) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Patients who have received a live vaccine within 30 days of the start date of the planned study therapy. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Has a known history of active TB (Bacillus Tuberculosis)
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 2 weeks of the first dose of treatment.
* Has had a prior chemotherapy, immunotherapy, biological therapy, targeted small molecule therapy, or radiation therapy within 3 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy, alopecia or hypothyroidism are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy events due to a previously administered agent.
* Presence of a gastrointestinal condition that may affect drug absorption
* Known allergy or reaction to any component of either study drug formulation
* Women who are pregnant or breast feeding
* Subjects expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment(s).
* Inability to comply with protocol required procedures
* Subjects receiving Monoamine Oxidase Inhibitors (MAOIs) or drug which has significant MAOI activity (meperidine, linezolid, methylene blue) within the 21 days before screening.
* Any history of Serotonin Syndrome (SS) after receiving serotonergic drugs.
* History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful. Screening QTc interval 480 milliseconds is excluded. In the event that a single QTc is ≥ 480 milliseconds, the subject may enroll if the average QTc for the 3 ECGs is < 480 milliseconds. For subjects with an intraventricular conduction delay (QRS interval > 120 milliseconds), the JTc interval may be used in place of the QTc with the approval of the principal investigator. The JTc must be < 340 milliseconds if JTc is used in place of the QTc. Subjects with left bundle branch block are excluded.

Note: QTc prolongation due to pacemaker may enroll if the JTc is normal.

* Use of any UGT1A9 inhibitor from screening through follow-up period, including the following: diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid.
* History of prior therapy with an IDO1 inhibitor in combination with an anti-PD-1/anti-PD-L1 agent/any other drug specifically targeting checkpoint pathways. Patients who have received prior therapy with single agent anti-PD-1/anti-PD-L1 therapy or single agent IDO1 inhibitor will be eligible for this study.
* Presence of any other concurrent active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D'Angelo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UPS, Liposarcoma or Pleomorphic Liposarcoma | Leiomyosarcoma | Vascular Sarcoma Subtypes | Other
Started | 10 | 5 | 5 | 10
Completed | 1 | 0 | 0 | 0
Not Completed | 9 | 5 | 5 | 10
Not completed — Adverse Event | 1 | 0 | 2 | 1
Not completed — Lack of Efficacy | 7 | 4 | 1 | 9
Not completed — Change in therapy | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UPS, Liposarcoma or Pleomorphic Liposarcoma | Leiomyosarcoma | Vascular Sarcoma Subtypes | Other | Total
Number analyzed (Participants) | 10 | 5 | 5 | 10 | 30
Age, Continuous [Median (Full Range); unit: years] | 54 [35 to 78] | 62 [37 to 76] | 53 [34 to 71] | 45 [24 to 75] | 54 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 4 | 12
  Male | 7 | 2 | 3 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 5 | 4 | 10 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 9 | 5 | 2 | 7 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 5 | 5 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Best Objective Response Rate
Description: by RECIST 1.1.
Time Frame: by 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | UPS, Liposarcoma or Pleomorphic Liposarcoma | Leiomyosarcoma | Vascular Sarcoma Subtypes | Other
Number analyzed (Participants) | 10 | 5 | 5 | 10
Participants
  Participants with PR | 0 | 1 | 0 | 0
  Participants without PR | 10 | 4 | 5 | 10

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | UPS, Liposarcoma or Pleomorphic Liposarcoma | Leiomyosarcoma | Vascular Sarcoma Subtypes | Other
All-Cause Mortality (participants affected / at risk) | 7/10 | 4/5 | 2/5 | 9/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/5 | 0/5 | 1/10
Other Adverse Events (participants affected / at risk) | 10/10 | 5/5 | 5/5 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UPS, Liposarcoma or Pleomorphic Liposarcoma (N=10) | Leiomyosarcoma (N=5) | Vascular Sarcoma Subtypes (N=5) | Other (N=10)
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Fever (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UPS, Liposarcoma or Pleomorphic Liposarcoma (N=10) | Leiomyosarcoma (N=5) | Vascular Sarcoma Subtypes (N=5) | Other (N=10)
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
BCC L eye (Eye disorders) | 0 | 0 | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 1 | 2
Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 3
Creatinine increased (Investigations) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 3
Early Satiety (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Edema face (General disorders) | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 3 | 0 | 1 | 1
Elevated ALK (Investigations) | 0 | 0 | 0 | 1
Elevated ALP (Investigations) | 0 | 1 | 0 | 0
Elevated AST (Investigations) | 0 | 0 | 0 | 1
Elevated Lipase (Investigations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Fatigue (General disorders) | 4 | 4 | 4 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Fever (General disorders) | 3 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 3 | 1 | 1 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 2 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 1 | 0
Localized edema (General disorders) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1
Lymphedema (Vascular disorders) | 0 | 1 | 0 | 0
Melena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 5 | 3 | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 2 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Periorbital (Eye disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 2
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Sensitivity of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Serum amylase increased (Investigations) | 2 | 0 | 2 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Skin changes to left temple (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Stye R eye (Eye disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Investigations) | 1 | 0 | 1 | 2
Thromboembolic Event (Vascular disorders) | 1 | 0 | 1 | 1
Thrush (Infections and infestations) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Weight gain (Investigations) | 1 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT03414229/Prot_SAP_000.pdf